CLINICAL TRIAL: NCT01153919
Title: A Double-Blind, Placebo-controlled Phase II Study to Assess the Efficacy and Safety of Romiplostim, Administered Once Weekly to Thrombocytopenic Hepatitis C (HCV) Infected Subjects Who Are Not Candidates for Antiviral Treatment With Pegylated Interferon and Ribavirin Due to Persistent Thrombocytopenia
Brief Title: Romiplostim in Treating Hepatitis C-Infected Patients With Thrombocytopenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Approval of several new agents for the treatment of HCV infection would mitigate the future need for interferon HCV treatment
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NC-HEM-07-5; NCI-2010-00358
Record Dates: First submitted 2010-06-24; First posted 2010-06-30 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis C Infection; Thrombocytopenia
MeSH Terms: conditions — Hepatitis C; Thrombocytopenia | interventions — romiplostim; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): Patients receive romiplostim subcutaneously once weekly for 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: romiplostim; Drug: ribavirin; Biological: PEG-interferon alfa-2a; Other: laboratory biomarker analysis
- Arm II (Placebo Comparator): Patients receive placebo subcutaneously once weekly for 8 weeks. Patients failing to achieve a platelet count of > 100,000/L cross over to arm I.
  Interventions: Drug: ribavirin; Other: placebo; Biological: PEG-interferon alfa-2a; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: romiplostim — Given subcutaneously
  Other Names: AMG 531; Amgen megakaryopoiesis protein 2; Nplate
  Arms: Arm I
Drug: ribavirin — Given orally
  Other Names: ICN-1229; Rebetol; RIBA; RTCA; Viramide; Virazole
Other: placebo — Given subcutaneously
  Other Names: PLCB
  Arms: Arm II
Biological: PEG-interferon alfa-2a — Given subcutaneously
  Other Names: PEG-IFNA2a; PEGASYS; pegylated interferon alfa-2a
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Romiplostim may cause the body to make platelets.

PURPOSE: This randomized phase II trial is studying how well romiplostim works in treating hepatitis C-infected patients with thrombocytopenia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the platelet count response to administration of weekly romiplostim patients with HCV infection whose initial platelet count is < 70,000/L.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of romiplostim the treatment of patients with HCV infection and thrombocytopenia; including physical symptoms and findings, hematologic, serum chemistries and liver function tests and adverse events.

II. To assess the ability of romiplostim to enable subjects to achieve a platelet count sufficient to start antiviral therapy.

III. To assess the ability of romiplostim to maintain platelet counts greater than 50,000/L while receiving antiviral therapy with pegylated interferon and ribavirin.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive romiplostim subcutaneously once weekly for 8 weeks in the absence of disease progression or unacceptable toxicity.

Arm II: Patients receive placebo subcutaneously once weekly for 8 weeks. Patients failing to achieve a platelet count of > 100,000/L cross over to arm I.

Patients achieving a platelet count of > 100,000/L at 8 weeks receive PEG-interferon alfa-2a subcutaneously once weekly and oral ribavirin once daily. Treatment repeats every 7 days for 24-48 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 and 36 weeks.

ELIGIBILITY:
Inclusion

* All patients with HCV virus infection documented by detectable plasma HCV antibodies and RNA who would be excluded by FDA criteria for antiviral treatment with peginterferon-alpha 2a and ribavirin due to thrombocytopenia (platelets < 70,000/L); patients cannot have received previous anti-viral therapy with interferon/ribavirin
* Liver biopsy indicating chronic hepatitis within the previous 2 years
* Mean platelet count of < 70,000/L on two repeated measurements in a two week screening period with no single count >= 75,000/L
* Neutrophil count of >= 1000/mcl
* Hemoglobin >= 11gm/dL and no evidence of active bleeding
* Prothrombin Time (PT) INR < 1.6 seconds
* Albumin >= 2.5 gm/dL
* ALT >= 1.2 and < 10 times upper limit of normal
* No evidence of either ischemic change or cardiac injury on 12-lead electrocardiogram (EKG)
* Negative pregnancy test and women must be using adequate contraception for at least 2 weeks prior to enrollment and while enrolled in the study
* Signed informed consent within 2 weeks of enrollment and randomization

Exclusion

* Received previous anti-viral therapy with interferon/ribavirin
* Child's Class B and C or acute decompensated liver disease
* Human Immunodeficiency Virus (HIV) infection or co-infected with hepatitis B virus
* Any untreated active infection
* Active malignancy, known primary bone marrow disorder (myelodysplasia, myeloproliferative disease, etc.), or history of blood or bone marrow transplantation; patients with documented hemoglobinopathies
* Active vasculitis associated with cryoglobulinemia as manifested by either renal disease or dermatologic findings
* Positive pregnancy test or men with pregnant partners
* Creatinine and BUN of greater than twice (2x) the upper limits of normal
* History of venous or arterial thrombosis, myocardial infarction or thrombotic stroke
* Patients who in the investigators opinion will fail to be compliant or have other contraindication to treatment on this study
* Other inherited or acquired liver disease
* Previous solid organ transplant
* Known hypersensitivity to E. coli derived recombinant proteins
* Active rheumatologic disease including Systemic Lupus Erythematosis
* Known history of Disseminated Intravascular Coagulation, Hemolytic Uremic Syndrome, or Thrombotic Thrombocytopenic Purpura

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-06-30 (Actual); Primary Completion 2014-07-14 (Actual); Study Completion 2018-07-14 (Estimated)

PRIMARY OUTCOMES:
Mean platelet count for actively treated and placebo treated subjects | Weeks 6-8

SECONDARY OUTCOMES:
Incidence of adverse events, including clinically significant changes in laboratory values and the incidence of antibody formation | Weeks 1-24
Number of subjects in each treatment group who achieve a platelet count of greater or equal to 100,000/L | Week 8
Number of patients originally receiving active treatment who maintain a platelet count > 50,000/L while receiving anti-viral therapy with pegylated interferon and ribavirin | Weeks 9-24
Changes in plasma HCV viral load during treatment with romiplostim alone | Weeks 1-8
Incidence of sustained viral response achieved during treatment with anti-viral therapy in combination with romiplostim | Weeks 9-24

CONTACTS AND LOCATIONS:
Overall Officials: Howard Liebman, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States